CLINICAL TRIAL: NCT02697864
Title: A Phase 1, Open-Label, Three Period Randomized, Single Dose Study To Estimate The Relative Bioavailability Of Pf-06291826 (Tafamidis) Free Acid Tablet Formulation Versus Commercial Capsule In Healthy Subjects Under Fasted Conditions
Brief Title: A Study Comparing Amounts of Tafamidis In The Blood Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461051; 2016-000295-16 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Healthy
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 48.8 mgA tafamidis free acid tablet (Experimental)
  Interventions: Drug: tafamidis
- 58 mgA tafamidis free acid tablet (Experimental)
  Interventions: Drug: tafamidis
- 4 soft gel capsules of 20 mg tafamidis meglumine (Experimental)
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis

SUMMARY:
3 different formulations and doses of tafamidis will be compared. Subjects will be fasted for each test and every subject will test all 3 different formulations. After swallowing tafamidis, tafamidis blood concentrations will be measured periodically for 6 days. After 14 days, subjects will take a different formulation of tafamidis and tafamidis blood concentrations will be measured periodically for 6 days. After another 14 days, the last formulation will be tested in the same way.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-child bearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 and total body weight more than 50 kg (110 lbs).

Exclusion Criteria:

* Blood pressure at screening visit of greater than 140 mm Hg (systolic) or 90 mg Hg (diastolic).
* Use of prescription or nonprescription drugs supplements within 7 days prior to 7 days of the study.
* Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time Curve (AUC) | 120 hours
Maximum Observed Plasma Concentration (Cmax) | 120 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 120 hours
Mean residence time (MRT) | 120 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 120 hours
Plasma Decay Half-Life (t1/2) | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461051&StudyName=A+Phase+1%2C+Open%E2%80%91label%2C+Three+Period+Randomized%2C+Single+Dose+Study+To+Estimate+The+Relative+Bioavailability+Of+Pf%E2%80%9106291826+%28tafamidis%29+Free+Acid+Tablet+Formulation+Versus+Commercial+Capsule+In+Healthy+Subjects+Under+Fasted+Conditions